CLINICAL TRIAL: NCT01031147
Title: Detection of Intracranial Aneurysm With Non-enhanced, Three-dimensional Time-of-flight Magnetic Resonance Angiography(3D-TOF-MRA): a Prospective Comparison With Three-dimensional Reconstructed Digital Subtraction Angiography (3D RDSA)
Brief Title: Contrast-free Magnetic Resonance Angiography (MRA) at 3.0 T for Intracranial Aneurysm Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Cerebral aneurysm study in China, The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University
Other Study IDs: CASC3
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2009-12

CONDITIONS: Intracranial Aneurysms
Keywords: Magnetic resonance angiography; Intracranial aneurysm; Digital subtraction angiography; Volume rendering
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Magnetic resonance angiography: Three-dimensional time-of-flight magnetic resonance angiography(3D-TOF-MRA) was used to detect the intracranial aneurysms in this study
  Interventions: Other: Examination

INTERVENTIONS:
Other: Examination — 3D-TOF-MRA was performed for suspected patients to detect intracranial aneurysm, and subsequently underwent digital subtraction angiography
  Other Names: 3D-TOF-MRA

SUMMARY:
The Chinese Cerebral Aneurysms Survey is a continuing prospective study to evaluate the effectiveness of unenhanced, three-dimensional time-of-flight magnetic resonance angiography (3D-TOF-MRA) with volume rendering (VR) at 3-T in the detection of intracranial aneurysms.

DETAILED DESCRIPTION:
Recent years,three-dimensional time-of-flight MRA (3D-TOF-MRA) has become a useful, contrast-free method for observing intracranial vessels and is widely utilized as a screening examination for intracranial aneurysms. The studies available in Medline show mixed results.Some of these studies just included MRI/MRA in the analysis, which have a high rate of false-positives and are unreliable, and some were lack of control (ruptured aneurysm), precise numbers of false-positive results, standard images process and review, or corroborative IADSA in some patients. Furthermore, most previous studies included small sample size with aneurysm detection at 0.5-T or 1.5-T MR. Thus, these results have been inconclusive because of certain pitfalls in these studies.

Since 2007, we have conducted a clinical study to objective detection of intracranial aneurysms in our routine diagnostic work-up of intracranial aneurysms by our neuroradiologists using a standard procedure with 3D-TOF-MRA with VR at 3T. The investigators want to establish the quality data to prospectively compare 3D-TOF-MRA with VR at 3T vs 3D-RDSA in the diagnosis of intracranial aneurysms in a largest cohort of patients and test it accuracy in screening for suspected patients

ELIGIBILITY:
Inclusion Criteria:

* Suspected or known intracranial aneurysms

Exclusion Criteria:

* Patient's inability to cooperate
* Chronic renal failure patients
* Any patients with a contraindication to MRA examination, such as pacemaker, orbital metallic foreign body, coronary stent, etc.
* Any patients with a contraindication to DSA examination, such as allergic to contrast medium, etc.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We estimated that a sample of 350 patients including 12% dropout rate would be enrolled to determine an accuracy of VR 3D-TOF-MRA versus VR RDSA as reference standard with a 95% confidence interval of 5% (i.e., a standard error of approximately 2.5 %) above and below the expected VR 3D-TOF-MRA accuracy of 95%. A P value of 0.05 was considered to indicate statistical significance.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated People's Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li MH, Cheng YS, Li YD, Fang C, Chen SW, Wang W, Hu DJ, Xu HW. Large-cohort comparison between three-dimensional time-of-flight magnetic resonance and rotational digital subtraction angiographies in intracranial aneurysm detection. Stroke. 2009 Sep;40(9):3127-9. doi: 10.1161/STROKEAHA.109.553800. Epub 2009 Jun 25. PMID 19556531